CLINICAL TRIAL: NCT07252063
Title: Assessment of Sensory Block Distribution and Postoperative Analgesia Following Ultrasound-Guided Interfascial Plane Blocks in Living Liver Donors: A Prospective Observational Study
Brief Title: Sensory Distribution and Postoperative Analgesia of Ultrasound-Guided Interfascial Plane Blocks in Living Liver Donors
Status: Recruiting | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Selma Basyigit, Department of Anesthesiology, Bahçeşehir University
Other Study IDs: Liver mapping
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: interfascial plane block — Ultrasound-guided interfascial plane blocks are administered at the end of surgery. Block selection and needle entry points are determined according to the surgical incision line and the location of abdominal drains. All blocks are performed under real-time ultrasound guidance using the institution's standardized protocol.
Other: patient controlled analgesia device — Intravenous patient-controlled analgesia is initiated in the postoperative period according to the institution's standard protocol. PCA settings, opioid type, basal infusion (if applicable), and bolus doses follow routine clinical practice and are recorded for analysis. PCA use during the first 24 hours is monitored to assess postoperative analgesic requirements.
Other: cutaneus sensory mapping — Cutaneous sensory mapping is performed in the post-anesthesia care unit (PACU) at the second postoperative hour. Sensory blockade is assessed using a standardized pinprick test applied radially from medial to lateral directions. The borders of the blocked and unblocked regions are marked on the skin using a UV-visible dermatographic pen. Mapping is conducted over the mid-abdominal and lateral abdominal regions, and the total cutaneous coverage areas are subsequently calculated for analysis.

SUMMARY:
Living liver donor hepatectomy at our institution routinely includes ultrasound-guided interfascial plane blocks as part of postoperative analgesia. Although these blocks have become increasingly used in donor hepatectomy, their cutaneous sensory distributions and block-related dermatomal coverage have not been systematically evaluated, with only anecdotal reports available in the literature.

This prospective observational study aims to assess both the sensory blockade patterns and the early postoperative analgesic performance of interfascial plane blocks administered to living liver donors. Following surgery, all consenting donors receive the institution's standard block protocol. Cutaneous sensory mapping is performed in the post-anesthesia care unit (PACU) at the second postoperative hour. Pain intensity and analgesic requirements within the first 24 hours are also recorded.

The study is designed to provide objective data on the dermatomal coverage and postoperative analgesic effects of contemporary ultrasound-guided interfascial plane blocks used in living liver donor surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult living liver donors undergoing elective donor hepatectomy

Age 18 to 65 years

ASA physical status I-II

Patients who have received ultrasound-guided interfascial plane blocks as part of their postoperative analgesia

Ability to cooperate with postoperative sensory mapping procedures

Patients who agree to participate and provide written informed consent

Exclusion Criteria:

Patients who refuse to participate or do not provide written informed consent

Patients who have not received any ultrasound-guided interfascial plane block

ASA physical status > II

Presence of surgical incisions or wound complications preventing reliable sensory mapping

Prior major abdominal surgery that may alter cutaneous innervation patterns

Cognitive impairment limiting the ability to cooperate with sensory testing

Known psychiatric disorders (e.g., major depression, mania, schizophrenia) that may interfere with postoperative assessment

Local infection, skin disease, or dermatologic condition preventing accurate cutaneous mapping

Allergy or contraindication to local anesthetics used in the block

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult living liver donors undergoing elective donor hepatectomy at a tertiary care center. All participants receive ultrasound-guided interfascial plane blocks as part of the institution's routine postoperative analgesia protocol. Eligible donors are aged 18 to 65 years, classified as ASA physical status I-II, and able to cooperate with postoperative cutaneous sensory mapping procedures. Individuals with contraindications to regional anesthesia, conditions preventing accurate sensory assessment, or those who decline participation are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous sensory block area mapping for different regional anesthesia techniques in liver donor surgery | At 120 minutes after block administration in the post-anesthesia care unit (PACU).
  The cutaneous sensory block area produced by the regional anesthesia technique will be evaluated at the 120th minute post-block using a standardized pinprick test. Sensory borders will be identified radially and marked on the skin with a UV-visible marker. Each mapped region will be photographed with a calibrated reference scale placed on the skin. These images will be processed using a predefined digital template to calculate the total blocked surface area in square centimeters. The resulting measurements will be used to characterize the sensory distribution of the interfascial plane blocks in living liver donors.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir Unişversity Medicalpark Goztepe hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No